CLINICAL TRIAL: NCT03386331
Title: The Influence of Vitamin D Receptor (VDR) Gene Polymorphisms (BsmI, TaqI, ApaI, FokI) on Weight Loss by Diet and Exercise Interventions in Non-diabetic Overweight and Obese Subjects
Brief Title: VDR Gene Polymorphisms and Weight Loss in Non-diabetic Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5/4/8-9/11/NCDII
Record Dates: First submitted 2017-07-26; First posted 2017-12-29 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet and Exercise (Other)
  Interventions: Behavioral: diet and exercise

INTERVENTIONS:
Behavioral: diet and exercise — Diet and lifestyle intervention

SUMMARY:
This is a six months intervention study in non-diabetic overweight and obese subjects. Subjects will be counseled for weight loss through diet and exercise. Diet and exercise will be recommended as per the regular norms for weight loss (weight loss ≥10% from baseline weight will be considered as a significant loss of weight) for overweight and obese subjects. A sample size of 90 subjects was calculated but assuming a drop out rate of 20%, 110 subjects will be enrolled. Enrolled subjects will be measured at every visit (monthly) for weight, body composition measures of abdominal obesity and skin folds. They would be assessed for compliance with diet and exercise. Detailed analysis of body composition including DXA, biochemical analysis will be performed at enrollment and after six months intervention. Statistical analysis will be performed to find association between measures of body composition for weight loss and genotypes of the VDR polymorphisms.

DETAILED DESCRIPTION:
This is a six months intervention study in non-diabetic overweight and obese subjects. Subjects will be counseled for weight loss through diet and exercise. Diet and exercise will be recommended as per the regular norms for weight loss (weight loss ≥10% from baseline weight will be considered as a significant loss of weight) for overweight and obese subjects. A sample size of 90 subjects was calculated but assuming a drop out rate of 20%, 110 subjects will be enrolled. Enrolled subjects will be measured at every visit (monthly) for weight, body composition measures of abdominal obesity and skin folds. They would be assessed for compliance with diet and exercise. Detailed analysis of body composition including DXA, biochemical analysis will be performed at enrollment and after six months intervention. Statistical analysis will be performed to find association between measures of body composition for weight loss and genotypes of the VDR polymorphisms.

VDR Polymorphisms

Polymorphisms in the VDR gene have been identified through out the complete VDR gene region and associated with cancer and autoimmune diseases. The FokI polymorphism is present in the translation site and results in the VDR protein being shortened by three amino acids and is not linked with any other VDR polymorphisms. This polymorphism predisposes to bone-disease, risk of cancer, immune mediated diseases 147-149,150, 151.

The common VDR gene polymorphisms are BsmI, TaqI, ApaI and FokI. These polymorphisms have shown varying results with insulin sensitivity and secretion.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 yrs
* BMI ≥ 23 kg/m2

Exclusion Criteria:

* Type 1 or Type 2 Diabetes.
* On drugs or meal supplements for weight loss.
* On calcium and or vitamin D supplement currently or in the previous six months.
* Have past or current history or family history of renal stones.
* Have participated in any other investigational drug study in the previous three months.
* Have any systemic diseases (cardiac, hepatic, endocrine or renal) or taking any kind of treatment more than one month in the last six months.
* Diagnosed malabsorption (celiac disease, Cohn's, ulcerative colitis) or history suggestive of malabsorption.
* Have past history of bariatric surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Body weight (Kg) | 6 months
  weight loss

SECONDARY OUTCOMES:
Genetic polymorphism | 6 months
  BsmI, TaqI, ApaI, FokI

CONTACTS AND LOCATIONS:
Locations (1):
- Anoop misra, New Delhi, India

IPD SHARING:
Plan to Share IPD: No